CLINICAL TRIAL: NCT05008068
Title: Effect of Local Application of Platelet-rich Fibrin Scaffold Loaded With Simvastatin on Peri-implant Bone Changes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Sara Fikry El Shafei, Principal investigator, British University In Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 0012490
Record Dates: First submitted 2021-08-02; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Platelet-rich Fibrin; Simvastatin
Keywords: Platelet-rich fibrin; Simvastatin; Bone loss; Peri-implant Bone Changes
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Each patient received two implants, one on each side of the arch. One side was treated with PRF alone and the other side with PRF +Simvastatin, at the time of Osteotomy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF alone (Experimental)
  Interventions: Drug: Simvastatin
- PRF in addition to Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin with PRF at site of osteotome

SUMMARY:
ACKGROUND: Simvastatin (SIM), a pharmacological drug used for hypercholesterolemia, has been found to have pleotropic effects on bones. Simvastatin together with the appropriate carrier may decrease bone loss around implants.

PURPOSE: To compare the long term effects of autologous PRF alone, and PRF loaded with SIM on peri-implant bone changes and implant stability in patients undergoing implant rehabilitation.

MATERIALS AND METHODS: A randomized controlled split-mouth studyincluding 8 males between the ages of 45-60 years. Each patient received two implants, one on each side of the arch. One side was treated with PRF alone and the other side with PRF +Simvastatin, at the time of Osteotomy. A cone-beam CT was used to evaluate bone changes around the insertion of implant sites atthree, six, and twelve months postoperatively. The secondary outcome included measuring implant stability using Ostell device at baseline and 3 months post insertion. To compare groups at different time periods, data was examined using a two-way (ANOVA) analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with a partially edentulous mandible indicated for rehabilitation with implant prostheses,
* any extractions, or surgeries performed at least six months earlier.

Exclusion Criteria:

* patients with systemic diseases affecting bone quality or resorption
* temporomandibular joint dysfunction,
* severe attrition or parafunctional habits,
* patients undergoing radiotherapy or chemotherapy,
* heavy smokers,
* vulnerable groups such as psychologically unstable patients

Ages: 45 Years to 60 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
The measurement of bone thickness | After 3 months of the osteotomy and application of Simvastatin
  Measuring unit in millimeters , measuring device is CBCT software
The measurement of bone thickness | After 6 months of the osteotomy and application of Simvastatin
  Measuring unit in millimeters , measuring device is CBCT software
The measurement of bone thickness | After 12 months of the osteotomy and application of Simvastatin
  Measuring unit in millimeters , measuring device is CBCT software

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in EGYPT, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No